CLINICAL TRIAL: NCT02958488
Title: Prospective Efficacy and Tolerance Data Collection in 34 to 36 Weeks Preterm Neonates Treated by High Flow Nasal Cannula for Respiratory Distress Syndrom
Brief Title: Efficacy and Tolerance of High Flow Nasal Cannula for Respiratory Distress Syndrom in Late Preterms (34-36 Weeks)
Acronym: PRIMAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9606
Record Dates: First submitted 2016-08-05; First posted 2016-11-08 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress Syndrom; High Flow Nasal Cannula
Keywords: 34 to 36 Weeks Preterm Neonates; Respiratory Distress Syndrom; High Flow Nasal Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preterm Neonates with Respiratory Distress Syndrome (Experimental): 34 to 36 Weeks Preterm Neonates with Respiratory Distress Syndrome
  Interventions: Device: High Flow Nasal Cannula

INTERVENTIONS:
Device: High Flow Nasal Cannula

SUMMARY:
The main objective of the study is to gather preliminary data on the effectiveness of High Flow Nasal canula (HFNC), provided since the delivery room, for ventilatory support in newborns of 34-36 weeks with moderate respiratory distress syndrome (RDS).

The secondary objective is to evaluate the safety of HFNC in this indication.

DETAILED DESCRIPTION:
Treatment with HFNC will start maximum 30 minutes after birth at an initial flow rate of 2L/Kg/min.

According to retraction signs, flow may be increased by gradual increments of 1L/min to reach a maximum flow rate of 5L/kg/minute.

Patients not improving after 2 hours of support with HFBNC will be hospitalized in the neonatal intensive care unit (NICU), and HFNC maintained as long as necessary, with regular attempts of weaning.

At any moment during the study, aggravation will lead to stop HFNC trial, and the infant management decided by the physician involved in the patient's care.

Aggravation is definined by one of the following conditions: Silverman-Anderson score > 6, and / or FiO2 > 0.5 and / or severe apneas and / or hemodynamic instability.

ELIGIBILITY:
Inclusion Criteria:

* Newborn premature between 34 and 36 weeks of gestational age
* Moderate RDS after 30 minutes of life while treated with + 5cm H2O positive airway pressure
* Presence of a dedicated pediatric nurse and pediatrician
* Parental consent

Exclusion Criteria:

* Need for early intubation
* Severe RDS, defined by one of the following: Silverman-Anderson score > 6, severe hypoxia (FiO2 > 0.5), hemodynamic disorders (HR> 180 / min, MABP <30mmHg, capillary refill time > 5s, pallor), and severe apneas (> 5s and / or with bradycardia <80 /min)
* 1 minute Apgar score < 3 and / or five minutes Apgar score < 7
* Birth weight < 1800g and / or IUGR <-2 SD
* Congenital heart, pulmonary, facial, or digestive malformation
* Subject not affiliated to social security system
* Legal representatives unable to understand the terms of the study

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Total duration of noninvasive ventilation | from the first minute of life to the end of the hospitalization in the Department of Neonatal Medicine of Montpellier University Hospital Center, i .e. usually up to a minimal corrected gestationnal age of 36 weeks.

SECONDARY OUTCOMES:
Rate of hospitalization in NICU for RDS | from the first minute of life to the end of the hospitalization in the Department of Neonatal Medicine of Montpellier University Hospital Center, i .e. usually up to a minimal corrected gestationnal age of 36 weeks.
Rate of RDS aggravation | from the first minute of life to the end of the hospitalization in the Department of Neonatal Medicine of Montpellier University Hospital Center, i .e. usually up to a minimal corrected gestationnal age of 36 weeks.
Rate of intubation | from the first minute of life to the end of the hospitalization in the Department of Neonatal Medicine of Montpellier University Hospital Center, i .e. usually up to a minimal corrected gestationnal age of 36 weeks.
Rate of good tolerance of LNHD technique | from the first minute of life to the end of the hospitalization in the Department of Neonatal Medicine of Montpellier University Hospital Center, i .e. usually up to a minimal corrected gestationnal age of 36 weeks.
Incidence of side effects, including pain and discomfort, skin lesions, abdominal distension, air leak syndrome, necrotizing enterocolitis, hypothermia, hypoglycemia | from the first minute of life to the end of the hospitalization in the Department of Neonatal Medicine of Montpellier University Hospital Center, i .e. usually up to a minimal corrected gestationnal age of 36 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Cambonie, Professor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided